CLINICAL TRIAL: NCT00302341
Title: International Randomized, Controlled Phase 3 Trial of DB289 Versus Trimethoprim-sulfamethoxazole for the Treatment of Acute Pneumocystis Jiroveci Pneumonia (PCP) in Patients With HIV/AIDS
Brief Title: DB289 Versus TMP-SMX for the Treatment of Acute Pneumocystis Jiroveci Pneumonia (PCP)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA Clinical Hold as of 12/21/07 due to safety concerns
Sponsor: Immtech Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C05-009
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Pneumonia, Interstitial Plasma Cell; Pneumocystis Carinii Pneumonia; Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Pulmonary disease; Dyspnea; Hypoxemia; AIDS; Pneumocystis jiroveci
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Lung Diseases; Dyspnea; Hypoxia; Acquired Immunodeficiency Syndrome | interventions — pafuramidine; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): pafuramidine maleate, oral tablet, 100 mg bid X 14 days
  Interventions: Drug: Pafuramidine maleate (DB289)
- 2 (Active Comparator): TMP/SMX oral tablet, 15 mg/kg, split tid X 21 days
  Interventions: Drug: Trimethoprim-Sulfamethoxazole (TMP-SMX)

INTERVENTIONS:
Drug: Pafuramidine maleate (DB289) — Oral tablet, 100 mg bid, 14 days
  Arms: 1
Drug: Trimethoprim-Sulfamethoxazole (TMP-SMX) — 15 mg/kg, oral tablet split tid X 21 days
  Other Names: Bactrim
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the non-inferiority of pafuramidine maleate (DB289)versus trimethoprim-sulfamethoxazole (TMP-SMX)for the treatment of mild to moderately severe Pneumocystis pneumonia (PCP).

DETAILED DESCRIPTION:
The gold standard treatment for PCP is trimethoprim-sulfamethoxazole (TMP-SMX). This drug is highly effective; however, a significant number of patients are unable to complete a course of therapy due to adverse events, some of which can be life-threatening. In addition, mutations that confer resistance to sulfa-based drugs in other microorganisms are increasingly being reported in P. jiroveci. A potential role of these mutations in conferring clinical resistance to PCP and in breakthroughs to prophylaxis regimens based on sulfa drugs is being actively studied. Second and third line agents or combinations for PCP treatment are also limited in efficacy and/or by adverse events.

A new agent such as pafuramidine maleate (DB289), which has well documented activity against P. carinii in animal models, documented efficacy in a preliminary study trial in HIV-infected patients with PCP that were intolerant or resistant to TMP-SMX, was well tolerated in this trial and demonstrated a low toxicity profile in Phase 1 studies, would meet a significant medical need. Furthermore, pafuramidine maleate is active against other pathogens responsible for significant morbidity and mortality in patients with AIDS in the developing world, like different strains of Plasmodium (malaria) and Cryptosporidium parvum. The decrease in the rate of PCP in countries where patients with AIDS have access to HAART will present a significant challenge to the completion of this development program. The last published trial of PCP treatment was conducted by the ACTG in 24 U.S. sites between May 1991 and june 1993. That study needed to decrease the planned sample size to 195 due to low enrollment. This represents an important challenge for our program.

ELIGIBILITY:
Inclusion Criteria:

* Documented or presumptive HIV infection
* Signs and symptoms of PCP present for at least 5 days
* Pneumocystis jiroveci confirmed in BAL fluid or induced sputum sample
* Suitable candidate for oral therapy
* Alveolar-arterial oxygen (A-a) gradient < or = 45 mm Hg on room air and partial pressure of oxygen (pO2) > or = 60 mm Hg
* No more than 48 hours of prior treatment in the preceding 7 days for PCP treatment at full doses; failure of Pneumocystis prophylaxis or use of medications recommended for treatment of PCP at doses less than recommended by the CDC Guidelines is acceptable.

Exclusion Criteria:

* Unwilling or unable to discontinue use of other medications with anti-PCP activity
* AIDS related cachexia (weight loss that is more than 10% of ideal body weight)
* Severe diarrhea and/or vomiting
* History of hypersensitivity or severe or life threatening toxicity to TMP-SMX, other sulfonamides or pentamidine
* Active illicit drug use
* Impending respiratory failure or need for intubation
* AST and ALT levels > 3 times the upper limit of normal
* History of pancreatitis
* Severe PCP
* Karnofsky score < or = 20
* Terminal HIV disease or life expectancy of less than 6 months
* Acute concurrent pulmonary pathological condition that would obscure the evaluation of response to therapy
* Concomitant use of amphotericin B, gangciclovir, cyclosporine, warfarin, thiazide diuretics, phenytoin, methotrexate, leucovorin
* Receipt of systemic corticosteroids (except replacement therapy) within 14 days of study entry at high doses for 3 or more consecutive days. Concomitant use of corticosteroids, other than replacement doses for adrenal insufficiency, is also excluded unless the patient meets the CDC criteria for use of corticosteroids for treatment of PCP
* Pregnant or lactating women
* The subject has been previously enrolled in the study

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the proportion of subjects with clinical success at the End of Treatment (Day 22) for the Modified Intent-to-Treat population (mITT). | Day 22

SECONDARY OUTCOMES:
The secondary efficacy endpoints will be the proportion of subjects with clinical success at the End of Treatment (Day 22)for the Per Protocol population and sustained clinical success at the End of Study (Day 42)in the Per Protocol and mITT populations. | Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Judith Aberg, MD, Principal Investigator — NYU School of Medicine; Preston Church, MD, Principal Investigator — Medical University of South Carolina; Laurence Huang, MD, Principal Investigator — University of California, San Francisco; Amanda Peppercorn, MD, Principal Investigator — UNC AIDS Clinical Trials- School of Medicine; Carl Fichtenbaum, MD, Principal Investigator — University of Cincinnati; Kathleen Mullane, DO, Principal Investigator — University of Chicago; Jose Vazquez, MD, Principal Investigator — Henry Ford Health Systems
Locations (7):
- United States (7):
  - University of California, San Francisco, California
  - The University of Chicago, Chicago, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - NYU School of Medicine, New York, New York
  - UNC AIDS Clinical Trials, Chapel Hill, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Medical University of SC, Charleston, South Carolina